CLINICAL TRIAL: NCT03125668
Title: Impact of Telephone Follow-up in Patient's Health-related Quality of Life During the First Six Months of Warfarin Use: Randomized Clinical Trial
Brief Title: Impact of Telephone Follow-up in Patient's Health-related Quality of Life That Use Warfarin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rafaela de Oliveira Manzato, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38736914.1.0000.5393
Record Dates: First submitted 2017-02-22; First posted 2017-04-24 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Quality of Life; Warfarin; Health Education; Patient Compliance
MeSH Terms: conditions — Health Education; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): At the hospitalization, patients receive the educational program (Power Point®Slides, booklets and orientation) about the use of warfarin. After hospital discharge they receive a telephone follow-up (five calls) and two Face to face counseling.
  Interventions: Behavioral: Educational Program; Behavioral: Telephone follow-up; Behavioral: Face to face counseling
- Control Group (Active Comparator): At the hospitalization, patients receive the educational program (Power Point®Slides, booklets and orientation) about the use of warfarin. After hospital discharge they receive two face to face counseling.
  Interventions: Behavioral: Educational Program; Behavioral: Face to face counseling

INTERVENTIONS:
Behavioral: Educational Program — At the hospitalization, patients receive the educational program with Power Point®Slides, booklets and orientation about the use of warfarin.
Behavioral: Telephone follow-up — After hospital discharge they receive a telephone follow-up (five calls for six months: 1st call in one week and the others calls month by month until six months).
  During the telephone calls the researcher talk with the patient about the topics that were approach in the educational intervention and motivate the patient to follow the recommendations for they have a successful treatment.
  Arms: Intervention Group
Behavioral: Face to face counseling — They receive two face to face counseling (1st meeting in three months and the 2nd meeting in six months after hospital discharge). In the face to face counseling the researcher collect the data about anxiety and depression again, health-related quality of life and adverse events related to oral anticoagulation therapy.

SUMMARY:
The purpose of this study is to test an educational program with telephone follow-up to improve health-related quality of life (HRQoL), treatment adherence, and reduce anxiety and depression symptoms in patients who are starting oral anticoagulants (OA).

DETAILED DESCRIPTION:
Randomized controlled trial (RCT) at two Brazilian public hospitals, one in Ribeirão Preto and another one in Américo Brasiliense, state of São Paulo, Brazil.

Both groups will receive the educational program (Power Point®Slides, booklets and orientation) at the hospitalization. After the hospital discharge, the intervention group will receive the telephone follow-up (five calls for six months: 1st call in one week and the others calls month by month until six months) and two face to face counseling (1st meeting in three months and the 2nd meeting in six months). The control group just receive the same face to face counseling (1st meeting in three months and the 2nd meeting in six months) after the hospital discharge.

The educational program consist in information about the use of Warfarin and approach the specific topics in Power Point®Slides: Physiology: Definition of oral anticoagulants, mechanisms of action and clinical indication; Medication: Dose, time, storage and duration of therapy; Monitoring: Meaning of International Normalized Ratio (INR) , collection period and doctor's appointments; Other medications: Drug interactions and those considered "natural"; Feeding: Eating foods rich in K vitamin and fats; Alcoholic beverage: Care about alcohol , and if it occurs, does not stop the Oral Anticoagulants; Gestation: Necessity to start IV anticoagulants; Activities: In physical, domestic or work activities to use protective measures; Health treatment: Warn about OA to other professional and take the card of INR values; Travels: On trips take the OA and be programmed to the realization of INR out of their units; Signs /Symptoms: Report underdose (thrombus formation) and overdose (bleeding), seek health care.

After the orientations with Power Point®Slides, the patients receive one booklet with the same informations and the researcher answer any questions that patients have about the anticoagulation therapy.

In this moment (at hospitalization) the researcher also collects the data about symptoms of anxiety and depression using the validated questionnaire.

During the telephone calls the researcher talk with the patient about the topics that were approach in the educational intervention and motivate the patient to follow the recommendations for they have a successful treatment.

In the face to face counseling (three and six months after hospital discharge) the researcher collect the data about anxiety and depression again, health-related quality of life and adverse events related to oral anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Both genders;
* To start the use of Warfarin for the first time during the current hospitalization;
* To have a phone.

Exclusion Criteria:

* To start the Oral Anticoagulation Therapy with another oral anticoagulant;
* To start the Warfarin for surgical procedures;
* To have visual or hearing impairments;
* Don't have cognitive conditions* to answer the questions of data collection instruments (measured by adapted questions from Pfiefer (1975);
* To have a cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Health-Related Quality of Life | Three and six months after hospital discharge
  The Duke Anticoagulation Satisfaction Scale (DASS) was developed by Samsa et al. (2004) and validated for the Brazilian population by Pelegrino et al. (2011). The scale have 25 items divided in three domains: Limitation (9 items); Hassles and burdens (8 items); Psychological Impacts (8 items). All items have seven response categories: "not at all", "a little", "somewhat", "moderately", "quite a bit", "a lot", and "very much". Possible range: 25 to 175 and lower scores, indicated better Health-Related Quality of Life.

SECONDARY OUTCOMES:
Change in Symptoms of Anxiety and Depression | At baseline, Three and six months after hospital discharge.
  The questionnaire "Hospital Anxiety and Depression Scale (HADS)" was developed by Zigmond and Snaith (1983) and validated and adapted to Portuguese by Botega et al. (1995). The HADS contains 14 multiple choice questions, divided into two subscales: anxiety and depression (composed of seven items each).This questionnaire will be used to collect the data at baseline and at six months.
Adherence | INR values during the six months follow-up
  Patient adherence to oral anticoagulation therapy will be assessed by the INR (International Normalized Ratio) stability that will be calculated by the percentage of time patients remain within the measurement range using the number of INRs within the therapeutic range, divided by the number of INRs collected.
Assessment and frequency of adverse events related to Warfarin | Three and six months after hospital discharge
  Three questions developed by the authors about adverse events related to Warfarin.

CONTACTS AND LOCATIONS:
Overall Officials: Rosana S Dantas, PhD, Study Chair — University of São Paulo at Ribeirão Preto College of Nursing
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No